CLINICAL TRIAL: NCT06331507
Title: Refinement and Assessment of New MRI Technologies for Cardiovascular Exams Using the Phillips Cardiac Magnetic Resonance (CMR) Patch
Brief Title: Refinement and Assessment of New MRI Technologies for Cardiovascular Exams Using the Phillips CMR Patch
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator choice
Sponsor: University of Michigan (Other)
Collaborators: Philips Health Care (Industry)
Responsible Party: Principal Investigator, Prachi P Agarwal, M.D., Clinical Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00176904
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CMR in CIED (Experimental): Patients at Michigan Medicine who come in for cardiac imaging procedures and who have CIEDs.
  Interventions: Device: CMR patch

INTERVENTIONS:
Device: CMR patch — The Cardiac Magnetic Resonance (MR) patch is a sequence modification for enhancing the images in patients with devices (CIED) for assessing heart muscle scar. The Philips tested patch supports multiple cardiac MR imaging enhancements compiled from several individual patches generated by multiple Philips MR research collaborators for use on 1.5 Tesla Philips scanners.

SUMMARY:
This study is being done to improve image quality and provide the collaborator with feedback on wide band imaging in patients with cardiac implantable electronic devices (CIED).

ELIGIBILITY:
Inclusion Criteria: have a clinically ordered cardiac MRI exam at University of Michigan -

Exclusion Criteria: pregnant; contraindication to MRI

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prachi Agarwal, MD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine - University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CMR in CIED
Started | 292
Completed | 292
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CMR in CIED
Number analyzed (Participants) | 292
Age, Customized [Count of Participants; unit: Participants]
  >18 years | 292
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data was not acquired for participants.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 292

OUTCOME MEASURES:

1. Primary Outcome: Scan Speed
Description: Scan speed is time required to set-up and run the new technique relative to the standard method.
Time Frame: During the procedure (up to 90 minutes)
Population: Scan speed was originally intended to be a form of feedback to the collaborator. Because of changes in standard practice and the patch sequence becoming mainstream, data was not collected for analysis.
Arm/Group | CMR in CIED
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: During procedure (up to 90 minutes)
Arm/Group | CMR in CIED
All-Cause Mortality (participants affected / at risk) | 0/292
Serious Adverse Events (participants affected / at risk) | 0/292
Other Adverse Events (participants affected / at risk) | 0/292

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT06331507/Prot_001.pdf